CLINICAL TRIAL: NCT07185165
Title: Eclipse: Flotufolastat F 18 to Determine Treatment Success Following Prostate Focal Therapy
Brief Title: An Investigational Scan (Flotufolastat F 18 PET/CT) for Detecting Residual or Recurrent Disease in Patients Who Completed Focal Therapy for Prostate Cancer.
Acronym: ECLIPSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-1371; NCI-2025-06280 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-09-05; First posted 2025-09-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (flotufolastat F-18 PET/CT) (Experimental): Patients receive flotufolastat F-18 IV. Then 50-100 minutes after injection, patients undergo whole-body PET/CT over 20-50 minutes. Patients then undergo PET/CT/ultrasound fusion biopsy within 3 months.
  Interventions: Procedure: Computed Tomography; Drug: Fluorine F 18 Flotufolastat; Procedure: Positron Emission Tomography; Procedure: Ultrasound-Guided Prostate Biopsy

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Fluorine F 18 Flotufolastat — Given IV
  Other Names: FLOTUFOLASTAT F-18; RHPSMA-7.3C
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Ultrasound-Guided Prostate Biopsy — Undergo PET/CT/ultrasound fusion biopsy

SUMMARY:
This phase II trial evaluates how well flotufolastat F 18 positron emission tomography (PET)/computed tomography (CT) imaging works to detect cancer that remains (residual) or that has come back (recurrent) after the completion of focal therapy for prostate cancer. Flotufolastat F 18 is a radioactive tracer that binds to prostate specific membrane antigen (PSMA), a protein over-expressed on prostate tumor cells. This allows for visualization of PSMA-expressing cells upon imaging. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of, in the case of this research, flotufolastat F 18. Because prostate cancer takes up flotufolastat F 18, it can be seen with PET. CT utilizes x-rays that track the body from the outside. CT images provide an exact outline of the organs and potential inflammatory tissue where it occurs in the body. The PET/CT scanner combines the PET and the CT scanners into a single device. This device combines the anatomic (body structure) information provided by the CT scan with the metabolic information obtained from the PET scan. Metabolic information means how much of the injected tracer is taken up by inflammatory tissue. Flotufolastat F 18 PET/CT imaging may be an effective and less invasive way to detect residual or recurrent disease in prostate cancer patients, compared to other methods.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the accuracy of fluorine F 18 flotufolastat (flotufolastat F 18) compared with prostate biopsy to determine treatment success following focal therapy of the prostate.

SECONDARY OBJECTIVE:

I. To evaluate the standard uptake volume (SUV) threshold of flotufolastat F 18 compared to Gleason score.

EXPLORATORY OBJECTIVE:

I. To compare how flotufolastat F 18 and gallium Ga 68 gozetotide (Ga 68 PSMA 11) are distributed within the prostate in men who have previously undergone focal therapy.

OUTLINE:

Patients receive flotufolastat F-18 intravenously (IV). Then 50-100 minutes after injection, patients undergo whole-body PET/CT over 20-50 minutes. Patients then undergo PET/CT/ultrasound fusion biopsy within 3 months.

After completion of study intervention, patients are followed up at 1 month post-biopsy and then every 12 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-90 at study enrollment
* History of prostate cancer
* Men who have had focal therapy (laser, cryotherapy, high-intensity focused ultrasound [HIFU], Tulsa Pro, irreversible electroporation [IRE], brachytherapy) within 6-36 months of enrollment

Exclusion Criteria:

* Contraindication to flotufolastat F 18 PET CT
* Contraindication to ultrasound-guided prostate biopsy
* Patients who are planned to have an x-ray contrast agent or other PET radiotracer < 24 hours prior to the PET scan
* Patients with castrate levels of testosterone secondary to androgen deprivation therapy
* Inability to provide written informed consent
* Known inability to remain still and lie flat for the duration of the PET/CT (about 30 minutes)
* Any investigational agents within 42 days prior to the day of the first dose
* Not able to understand and to follow study instructions and requirements. This also includes the inability to complete the study imaging and or biopsy procedures due to any reason (e.g., severe claustrophobia, inability to lie still for the entire imaging time, any condition that precludes raised arms position)

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2035-10-25 (Estimated); Study Completion 2036-10-25 (Estimated)

PRIMARY OUTCOMES:
Accuracy of fluorine F 18 flotufolastat (flotufolastat F 18) positron emission tomography (PET)/computed tomography (CT) in detecting residual or recurrent prostate cancer lesions | Up to 10 years

SECONDARY OUTCOMES:
Optimal standardized uptake value (SUV) threshold of flotufolastat F 18 PET/CT | Up to 10 years
  Will establish the optimal SUV threshold of flotufolastat F 18 PET/CT that correlates with the Gleason score obtained from prostate biopsies, establishing a quantitative imaging biomarker for assessing focal therapy success.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Brisbane, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States